CLINICAL TRIAL: NCT01463826
Title: Association Between Respiratory Problem and Dental Caries in Children With Bruxism
Brief Title: Respiratory Problems and Caries in Children With Bruxism
Acronym: RPCB
Status: Completed | Type: Observational
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Lara Jansiski Motta, PhD, University of Nove de Julho
Other Study IDs: br82622/08
Record Dates: First submitted 2011-10-28; First posted 2011-11-02 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Bruxism; Dental Caries
Keywords: bruxism; children; oral breathing; dental caries
MeSH Terms: conditions — Bruxism; Dental Caries

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children with bruxism: 14 children with bruxism
- children without bruxism: 19 children without bruxism

SUMMARY:
The aim of the present study are to determine whether there is an association between respiratory problems and dental caries in children who exhibit the habit of bruxism.

DETAILED DESCRIPTION:
Objectives: The aim of the present study was to determine whether there is an association between respiratory problems and dental caries in children who exhibit the habit of bruxism.

Method: Patient histories were taken and clinical exams were performed on 90 children for selection and allocation to one of two groups. For the determination of bruxism, a questionnaire was administered to parents/guardians and an oral clinical exam was performed based on the criteria of the American Academy of Sleep Medicine. Thirty-three male and female children between four and seven years of age participated in the present study - 14 children with bruxism and 19 children without bruxism. The data were statistically analyzed using the chi-square test, with level of significance set at 5% (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Children with either the complete primary or mixed dentition who were not in dental treatment

Exclusion Criteria:

* Children in dental treatment

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with either the complete primary or mixed dentition who were not in dental treatment were included in the study and divided into two groups: those with bruxism and those without bruxism. For the diagnosis of bruxism, a questionnaire was administered to determine the occurrence of teeth clenching/grinding and a physical exam was performed for the determination of dental wear based on the criteria of the American Academy of Sleep Medicine. Dental caries were determined based on the criteria of the World Health Organization
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Motta, PhD, Principal Investigator — Nove de Julho University